CLINICAL TRIAL: NCT07247526
Title: The Effect of Preoperative Hot Water Foot Bath on Anxiety Level and Physiological Parameters in Patients With Pituitary Adenoma
Brief Title: Effect of Foot Bath on Anxiety and Physiological Parameters
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Seher Ünver, Professor Dr., Trakya University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2024/10
Record Dates: First submitted 2025-07-31; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Pituitary Adenoma; Surgery
Keywords: foot; physiological parameters; anxiety
MeSH Terms: conditions — Pituitary Neoplasms; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Experimental: Intervention Group Participants in this study group will be asked to keep their feet in hot water at 40oC (40 degrees Celsius) for 20 minutes, 1 hour before the surgery, on the day of surgery.
  Intervention: Other: Hot water foot bath No Intervention: Control Group Participants in this study group will receive standard service clinic procedure and will not receive a hot water foot bath.
Who Masked: Outcomes Assessor
Masking Description: The data analysed by a independent researcher
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants in this study group will be asked to keep their feet in hot water at 40oC (40 degrees Celsius) for 20 minutes, 1 hour before the surgery, on the day of surgery.
  Interventions: Other: Hot water foot bath
- Control Group (No Intervention): Control Group Participants in this study group will receive standard service clinic procedure and will not receive a hot water foot bath.

INTERVENTIONS:
Other: Hot water foot bath — Keeping feet in 40oC (40 Degrees Celsius) hot water for 20 minutes
  Arms: Intervention Group

SUMMARY:
The aim of this study is to examine the effect of hot water foot bath applied before pituitary adenoma surgery on anxiety level and physiological parameters. The main hypotheses are:

* H1: Foot bath applied before surgery reduces the state anxiety level of patients.
* H01: There is no difference between the preoperative mean arterial pressure of the patients in the foot bath applied study group and the control group.
* H02: There is no difference between the preoperative heart rate of the patients in the foot bath applied study group and the control group.
* H03: There is no difference between the preoperative respiratory rates of the patients in the foot bath applied study group and the control group.
* H04: There is no difference between the preoperative body temperatures of the patients in the foot bath applied study group and the control group.
* H05: There is no difference between the preoperative oxygen saturations of the patients in the foot bath applied study group and the control group.
* H06: There is no difference between the preoperative pain levels of the patients in the study group and the control group where foot bath was applied.

On the day of surgery, participants will be asked to keep their feet in 40 hot water for 20 minutes, 1 hour before the surgery.

If there is a comparison group: Researchers will compare the control group to see if there are any differences in the patients' anxiety level and physiological parameters.

DETAILED DESCRIPTION:
Group allocation of the patients was done through using Random Allocation Software program and patients were allocated into two groups: the intervention group and the control group.

The study was planned in three stages. In the first stage, the researcher nurse visited the patients in the study and control groups, who had been admitted to the ward at least 1 day before the surgery and who would be transferred to the operating room within 1 hour, in the single-person ward room, and after explaining the purpose of the research, she obtained the verbal and written consent of the patients who agreed to participate in the research. The Patient Information Form was filled out by the researcher nurse and the patients' state and trait anxiety levels were evaluated using STAI. The physiological parameters of the patients were evaluated by another nurse working in the ward due to the single-blind application of the study, and the results were recorded in the 0th minute section of the Patient Monitoring Table. Patients' pain levels were evaluated with VAS and anxiety levels with VAS-A. For this purpose, patients were asked to mark their scores on the scale.

In the second stage, the patients in the study group were asked to stand in a sitting position on the edge of the bed with their feet hanging down. The tub of the device to be used in the hot water foot bath was filled with water to cover 4-5 fingers above the patient's ankles and the temperature was adjusted to 40°C. Patients were asked to soak their feet in water for 20 minutes. During the intervention period, the researcher nurse was in the opposite room to monitor sudden changes in the patient's condition. After 20 minutes, the patients were asked to take their feet out of the water and were allowed to dry their feet by wrapping a towel around them. Patients in the control group were asked to remain in a comfortable sitting position for 20 minutes and were allowed to rest. The patients did not undergo any procedure.

In the third stage, the state anxiety levels and physiological parameters of the patients in the study and control groups were evaluated by another nurse working in the ward due to the single-blind conduct of the research. The measurement results of physiological parameters were recorded in the 20th minute section of the Patient Monitoring Table in accordance with the group to which the patient belonged. Patients' pain levels were evaluated with VAS and anxiety levels with VAS-A. For this purpose, patients were asked to mark their scores on the scale. Trait anxiety level was not re-evaluated because it did not show any immediate change.

ELIGIBILITY:
Inclusion Criteria:

* Those who are over 18 years old,
* Having a caregiver with him/her,
* Those who will undergo elective pituitary adenoma surgery,
* Those who were hospitalized at least one day before their surgery,
* No known psychological problems,
* Conscious, oriented and able to communicate verbally,
* No known peripheral vascular disease,
* Not having diabetes,
* No open wounds on their feet,
* Staying in a single room,
* Patients who want to take a foot bath in 40 °C water

Exclusion Criteria:

* Those who are under 18 years of age,
* Without a caregiver,
* Not undergoing elective pituitary adenoma surgery,
* Not hospitalized at least one day before the surgery,
* Having a known psychological problem,
* Conscious, oriented and unable to communicate verbally,
* Known peripheral vascular disease,
* Having diabetes,
* Having open wounds on their feet,
* Staying in a double room,
* Patients who do not want to take a foot bath in 40 °C water

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Anxiety Level | On the day of surgery, 1 hour before surgery
  It will be evaluated using STAI (State-Trait Anxiety Inventory) and VAS-A (Visual Analog Scale-Anxiety). STAI: Scores between 0-19 indicate no anxiety, scores between 20-39 indicate mild anxiety, scores between 40-59 indicate moderate anxiety, scores between 60-79 indicate severe anxiety, and scores of 80 and above indicate panic-level anxiety. VAS-A shows the level of anxiety between the score of "0-no anxiety" and the score of "10-I feel a lot of anxiety".
Systolic and diastolic blood pressure | On the day of surgery, 1 hour before surgery
  Using an automatic measuring device, patients' systolic and diastolic blood pressure will be measured.
heart rate | On the day of surgery, 1 hour before surgery
  Using an automatic measuring device patients' heart rate will be measured.
respiratory rate | On the day of surgery, 1 hour before surgery
  Using an automatic measuring device, patients' respiratory rate will be measured.
body temperature | On the day of surgery, 1 hour before surgery
  Using an automatic measuring device, patients' body temperature will be measured.
oxygen saturation | On the day of surgery, 1 hour before surgery
  Using an automatic measuring device, patients' oxygen saturation will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Seher Ünver, Assoc. Prof., Principal Investigator — Trakya University; Ülkü Çolakoğlu, BSN, Principal Investigator — Trakya University
Locations (1):
- Seher Ünver, Edirne, Edirne, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No